CLINICAL TRIAL: NCT05509686
Title: The Immediate Effects of Intermittent Theta Burst Stimulation on Intracortical Excitability of the Primary Motor Cortex in Patients With Chronic Stroke: A Concurrent TMS-EEG Sham-controlled Crossover Study
Brief Title: The Immediate Effects of Intermittent Theta Burst Stimulation on Intracortical Excitability of the Primary Motor Cortex in Patients With Chronic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Kenneth N. K. Fong, Professor in Rehabilitation Sciences, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20200621001
Record Dates: First submitted 2022-08-18; First posted 2022-08-22 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Stroke
Keywords: stroke; theta burst stimulation; transcranial magnetic stimulation-evoked potentials; intracortical inhibition; cortical excitability
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A single-session intermittent theta burst stimulation (iTBS) (Experimental): The classical 600-pulse iTBS protocol is delivered to the motor hotspot over the ipsilesional hemisphere.
  Interventions: Device: Intermittent theta burst stimulation (iTBS)
- A single-session sham intermittent theta burst stimulation (iTBS) (Sham Comparator): The sham stimulation is the same as that of iTBS, but the coil is placed five centimeters away from the scalp.
  Interventions: Device: Sham intermittent theta burst stimulation (iTBS)

INTERVENTIONS:
Device: Intermittent theta burst stimulation (iTBS) — A single-session standard 600-pulse intermittent theta burst stimulation (iTBS) is applied to the ipsilesional primary motor cortex.
  Arms: A single-session intermittent theta burst stimulation (iTBS)
Device: Sham intermittent theta burst stimulation (iTBS) — The sham stimulation is the same as that of iTBS, but the coil is placed five centimeters away from the scalp. Electrical field simulation shows that the setups for sham stimulation would not induce any valid cortical activation.
  Arms: A single-session sham intermittent theta burst stimulation (iTBS)

SUMMARY:
This study is to investigate the immediate effects of intermittent theta burst stimulation (iTBS) on intracortical excitatory and inhibitory circuits, neural connectivity, and network properties in patients with chronic stroke, using transcranial magnetic stimulation and electroencephalogram (TMS-EEG) and TMS-electromyography (EMG) and approaches.

DETAILED DESCRIPTION:
The neurophysiological effect of intermittent theta burst stimulation (iTBS) has been examined with TMS-electromyography (EMG)-based outcomes in healthy people; however, its effects in intracortical excitability and inhibition are largely unknown in patients with stroke. Concurrent transcranial magnetic stimulation and electroencephalogram (TMS-EEG) recording can be used to investigate both intracortical excitatory and inhibitory circuits of the primary motor cortex (M1) and the property of brain networks.

This study is to investigate the immediate effects of iTBS on intracortical excitatory and inhibitory circuits, neural connectivity, and network properties in patients with chronic stroke, using TMS-EEG and TMS-EMG approaches.

In this randomized, sham-controlled, crossover study, 21 patients with chronic stroke receive two separate stimulation conditions: a single-session iTBS or sham stimulation applied to the ipsilesional M1, in two separate visits, with a washout period of five to seven days between the two visits after crossover. A battery of TMS-EMG and TMS-EEG measurements are taken before and immediately after stimulation during the visit.

ELIGIBILITY:
Inclusion Criteria:

1. suffered from first-ever, ischemic or hemorrhagic, unilateral stroke, verified by neuroimaging examinations such as CT or MRI.
2. detectable motor evoked potentials from the affected first dorsal interosseous muscle;
3. provided written informed consent.

Exclusion Criteria:

1. had any contraindication to transcranial magnetic stimulation;
2. had a known neurological disease excluding stroke, or psychiatric disease;
3. were using a psychostimulant, sedative, antidepressant, or antiepileptic medication.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Transcranial magnetic stimulation-evoked potential | Baseline (before iTBS stimulation)
  Single pulses evoked an initial response in electroencephalogram, followed by a series of time- and phase-locked positive and negative deflections which could spread to the connected brain areas. The evoked potential is called transcranial magnetic stimulation-evoked potential.
Transcranial magnetic stimulation-evoked potential | 10 minutes after a single-session iTBS stimulation
  Single pulses evoked an initial response in electroencephalogram, followed by a series of time- and phase-locked positive and negative deflections which could spread to the connected brain areas. The evoked potential is called transcranial magnetic stimulation-evoked potential.
Motor evoked potential (MEP) | Baseline (before iTBS stimulation)
  Single TMS pulses with suprathreshold intensity (120% of resting motor threshold of the stimulated cortex) applied to the primary motor cortex (M1) can produce recordable MEPs in contralateral muscles; additionally, the peak-to-peak amplitude of MEPs can be used to represent the corticospinal excitability
Motor evoked potential (MEP) | 10 minutes after a single-session iTBS stimulation
  Single TMS pulses with suprathreshold intensity (120% of resting motor threshold of the stimulated cortex) applied to the primary motor cortex (M1) can produce recordable MEPs in contralateral muscles; additionally, the peak-to-peak amplitude of MEPs can be used to represent the corticospinal excitability

SECONDARY OUTCOMES:
Cortical silent period | Baseline (before iTBS stimulation)
  The cortical silent period (cSP) is a protocol measuring the intracortical inhibition, in which suprathreshold test pulses (120% of resting motor threshold of the stimulated cortex) are applied to the contralateral M1, while participants sustain 30% maximum voluntary contraction. Specifically, cSP refers to the interruption of background electromyographic (EMG) activity after the TMS pulse.
Cortical silent period | 10 minutes after a single-session iTBS stimulation
  The cortical silent period (cSP) is a protocol measuring the intracortical inhibition, in which suprathreshold test pulses (120% of resting motor threshold of the stimulated cortex) are applied to the contralateral M1, while participants sustain 30% maximum voluntary contraction. Specifically, cSP refers to the interruption of background electromyographic (EMG) activity after the TMS pulse.
Short-interval intracortical inhibition | Baseline (before iTBS stimulation)
  Short-interval intracortical inhibition (SICI) is a form of paired-pulse protocol, in which a subthreshold conditioning pulse is delivered 2 ms before a suprathreshold test pulse. Theoretically, the amplitude of motor-evoked potentials (MEPs) evoked by a test pulse at a given intensity is suppressed compared with that evoked by a single pulse at the same intensity. Eight trials are recorded, with inter-trial intervals ranging from 4 s to 5 s. The intensity of test pulses is fixed at 120% of the resting motor threshold, and the intensity of the conditioning pulse is set at 80% of the resting motor threshold. The result of SICI is expressed as the ratio of a paired-pulse MEP amplitude to a single-pulse MEP amplitude.
Short-interval intracortical inhibition | 10 minutes after a single-session iTBS stimulation
  Short-interval intracortical inhibition (SICI) is a form of paired-pulse protocol, in which a subthreshold conditioning pulse is delivered 2 ms before a suprathreshold test pulse. Theoretically, the amplitude of motor-evoked potentials (MEPs) evoked by a test pulse at a given intensity is suppressed compared with that evoked by a single pulse at the same intensity. Eight trials are recorded, with inter-trial intervals ranging from 4 s to 5 s. The intensity of test pulses is fixed at 120% of the resting motor threshold, and the intensity of the conditioning pulse is set at 80% of the resting motor threshold. The result of SICI is expressed as the ratio of a paired-pulse MEP amplitude to a single-pulse MEP amplitude.
Intracortical facilitation | Baseline (before iTBS stimulation)
  The setups for the intensity of intracortical facilitation (ICF) are almost the same as those for SICI; however, the interstimulus interval is longer, 10 ms. Eight trials are recorded, with inter-trial intervals ranging from 4 s to 5 s. The intensity of test pulses is fixed at 120% of the resting motor threshold, and the intensity of the conditioning pulse is set at 80% of the resting motor threshold. The result of ICF is expressed as the ratio of a paired-pulse MEP amplitude to a single-pulse MEP amplitude.
Intracortical facilitation | 10 minutes after a single-session iTBS stimulation
  The setups for the intensity of intracortical facilitation (ICF) are almost the same as those for SICI; however, the interstimulus interval is longer, 10 ms. Eight trials are recorded, with inter-trial intervals ranging from 4 s to 5 s. The intensity of test pulses is fixed at 120% of the resting motor threshold, and the intensity of the conditioning pulse is set at 80% of the resting motor threshold. The result of ICF is expressed as the ratio of a paired-pulse MEP amplitude to a single-pulse MEP amplitude.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Fong, PhD, Principal Investigator — Hong Kong Polytechnic University, QT517, Hung Hom
Locations (1):
- Kenneth FONG, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
The data will be shared for research purpose upon reasonable request.